CLINICAL TRIAL: NCT05648578
Title: The Effect of Reiki Practice on Stress and Anxiety Levels in Nurses: A Randomized Controlled Trial
Brief Title: The Effect of Reiki Application on Stress and Anxiety Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Siirt University (Other)
Responsible Party: Principal Investigator, Zeliha Buyukbayram, Principal Investigator, Siirt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Siirt University
Record Dates: First submitted 2022-11-30; First posted 2022-12-13 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Stress
Keywords: Anxiety; Nursing; Reiki; Perceived stress
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Participants received reiki application for 4 weeks.
  Interventions: Other: Reiki attempt
- Control (No Intervention): No intervention was applied to the participants in the control group

INTERVENTIONS:
Other: Reiki attempt — Four reiki sessions were applied twice a week, on the same days of the week, lasting 25-35 minutes each.
  Arms: Experimental

SUMMARY:
The aim of this study is to determine the effect of reiki practice on stress and anxiety levels in nurses.

DETAILED DESCRIPTION:
It was a randomized controlled trial. Reiki was applied to the participants in the experimental group twice a week for two weeks. No intervention was applied to the participants in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer nurses were included in the research

Exclusion Criteria:

* Nurses, who had previous reiki experience and did not agree to participate in the study, were excluded

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Introductory Questionnaire | Baseline
  The introductory questionnaire created for descriptive expressions This questionnaire was prepared by the researchers in line with the literature and comprised questions about the age, gender, marital status, education level, unit, length of work, and job satisfaction of patients.
Perceived Stress Scale | Change from Baseline Stress at 2 week
  This scale used to measure perceived stress. Perceived stress scale was used to determine the stress of the participants. The scale is a 5-point Likert-type scale, ranging from "never (0)" to "very often (4)". The scale consists of 2 subscales: low self-esteem perception (items 4, 5, 6, 8, 9, 10, 13) and stress/discomfort perception (1, 2, 3, 7, 11, 12, 14). The total score on the scale ranges from 0 to 56. The high score indicates the excess of the individual perception of stress.
Beck Anxiety Inventory | Change from Baseline Anxiety at 2 week
  This scale used to determine the level of anxiety Beck Anxiety Inventory was used to determine the anxiety of the participants. The scale consists of 21 items. It is a 4-point Likert-type scale and includes "not at all", "mildly", "moderately", and "severely" options. It is in the range of 0-63 points, 8-15 points indicate low stress, 16-25 points moderate, and 26-63 points indicate high anxiety. A high score implies an excess of perception of stress by individuals.

CONTACTS AND LOCATIONS:
Locations (1):
- Siirt University, Siirt, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No